CLINICAL TRIAL: NCT00887692
Title: Comparison of Set-up Reproducibility Between Prone and Supine Intensity Modulated Radiotherapy (IMRT) for the Adjuvant Treatment of Breast Carcinoma After Lumpectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Wilfried De Neve, University Hospital Ghent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009/185
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Prone Position; Supine Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: prone and supine position — patients will be treated alternating daily between prone and supine position for breast radiotherapy.

SUMMARY:
10 patients will be treated alternating daily between prone and supine position for breast radiotherapy to compare set-up accuracy. Prone treatment will be given on the odds days and supine treatment on the even days.

ELIGIBILITY:
Inclusion Criteria:

* female patients
* multidisciplinary decision of adjuvant radiotherapy after lumpectomy for breast cancer
* minimum 18 years
* informed consent obtained, signed and dated before specific protocol procedures.

Exclusion Criteria:

* mastectomy
* need for axillary irradiation
* bilateral breast irradiation
* previous irradiation at the same time
* pregnant or breastfeeding
* mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study.
* patient unlikely to comply with the protocol; i.e. uncooperative attitude, inability to return for follow-up visits, and unlikely to complete the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Random set-up error | daily during radiotherapy

SECONDARY OUTCOMES:
Systemic set-up error | daily during radiotherapy
Respiration-related motion amplitude
time of treatment delivery | daily during radiotherapy
Dose-volume parameters | of planning

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Neve, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website of the University Hospital Ghent — http://www.uzgent.be